CLINICAL TRIAL: NCT05403190
Title: The Performance of da Vinci SP System on Extraperitoneal Approach Radical Prostatectomy-a Single Arm Pivotal Trial Initiated by Chang Gung Memorial Hospital, Taiwan
Brief Title: The Performance of da Vinci SP System on Extraperitoneal Approach Radical Prostatectomy
Acronym: CGMH-SPEAR-P
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Collaborators: Intuitive Surgical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 202101419A0C601
Record Dates: First submitted 2022-05-18; First posted 2022-06-03 (Actual); Last update posted 2023-02-22 (Actual); Status verified 2022-04

CONDITIONS: Prostate Cancer
Keywords: prostate cancer; radical prostatectomy; da Vinci SP system; extraperitoneal approach
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Study arm (Experimental): Patients with prostate cancer
  Interventions: Device: da Vinci SP system

INTERVENTIONS:
Device: da Vinci SP system — using da Vinci SP system to perform extraperitoneal approach radical prostatectomy

SUMMARY:
The objective of this study is to evaluate the performance and safety of da Vinci Single Port (SP) system on the surgery for extraperitoneal approach radical prostatectomy

DETAILED DESCRIPTION:
Enrolled subjects would receive extraperitoneal approach radical prostatectomy using da Vinci SP system and be assessed at baseline (preoperatively), during hospitalization, and postoperatively (at 1 month +/-4 days, 3 month +/- 7 days, 6 months +/- 10 days, 12month +/-14 days). The preoperative assessment includes any diagnostic tests to confirm the subjects' cancer status and eligibility for the intervention under consideration such as transrectal or transperineal biopsy, image studies for staging including MRI/CT and bone scan, and cardiopulmonary tests to evaluate risks for anesthesia. The hospitalization assessment includes the collection of perioperative and postoperative details, conversions, and complications. The postoperative assessment includes regular follow up studies to evaluate cancer status and functional outcome (For sexual function, the International Index of Erectile Function (IIEF-5) would be recorded before and after the surgery. For continence, the number of pads per day and 24hr total weight of pads would be recorded. No pad used or one safe pad per day with net wet ≤ 50gm would be considered as continent. International Prostate Symptom Score (IPSS) wound be recorded before and after the surgery to access voiding function).

ELIGIBILITY:
Inclusion Criteria:

1. Patients with biopsy-proved prostate cancer
2. Stage clinical T1-T2N0M0
3. Prostate volume ≦ 70cm (by transrectal ultrasound or other image studies)
4. BMI ≦ 35 kg/m
5. Low priority of nerve sparing (pre-op sexual dysfunction or don't care about sexual function)
6. Age between 18 and 78 years old
7. Suitable for minimally invasive surgery
8. Patients willing and able to provide informed consent
9. Patients willing and able to comply with study protocol requirements and follow-up

Exclusion Criteria:

1. Previous abdominal or pelvic major operation history
2. Previous radiation treatment to the pelvic area
3. Patients received transurethral resection of prostate in three months
4. Severe concomitant illness that drastically shortens life expectancy or increases risk of therapeutic interventions

   * Severe heart disease (NYHA functional class III-IV)
   * Severe lung disease (GOLD Group C-D)
5. Anatomy unsuitable for endoscopic visualization or minimally invasive surgery
6. Hemodynamic or respiratory instability after anesthesia
7. Working space restriction (e.g. kyphosis or severe scoliosis)
8. Emergency surgery
9. Untreated active infection
10. vulnerable populations

Ages: 18 Years to 78 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2023-07-31 (Estimated); Study Completion 2023-11-30 (Estimated)

PRIMARY OUTCOMES:
Success rate (%) | immediately after the surgery
  Percentage of successful extraperitoneal approach radical prostatectomy with da Vinci SP system (no conversion to conventional laparoscopic, multiport da Vinci surgery or open surgery; addition of access port to complete the procedure would not be considered as conversion.)

SECONDARY OUTCOMES:
Perioperative parameters-incision length (cm) | immediately after the surgery
  incision length
Perioperative parameters-console time (minutes) | immediately after the surgery
  console time
Perioperative parameters-blood loss (ml) | immediately after the surgery
  blood loss
Perioperative parameters-blood transfusion type | immediately after the surgery
  blood transfusion type
Perioperative parameters-blood transfusion unit | immediately after the surgery
  blood transfusion unit
Perioperative parameters-intra-operative complications (SATAVA system) | immediately after the surgery
  intra-operative complications accessed with SATAVA system, Grade 1 to 3, higher grade indicates serious complications
Perioperative parameters-oxidative stress | immediately after the surgery
  oxidative stress measured by the arterial malondialdehyde (MDA) level (micromole/L)
Postoperative parameters-length of hospital stay (days) | immediately after discharge (assessed up to 10 days)
  length of hospital stay
Postoperative parameters-pain scale (VAS score) | Every day during admission after the surgery (up to 7 days)
  pain scale accessed with visual analog scale (VAS) score, 1-10, higher score indicates more pain
Postoperative parameters-analgesic type | Every day during admission after the surgery (up to 7 days)
  analgesic type
Postoperative parameters-analgesic dose | Every day during admission after the surgery (up to 7 days)
  analgesic dose
Postoperative parameters-postoperative complications (CLAVIEN-DINDO system) | During admission after the surgery (up to 10 days)
  postoperative complications accessed with CLAVIEN-DINDO system, Grade I to V, higher grade indicates severe complications
Postoperative parameters-readmission and reoperation | If happens, on the day of re-admission or reoperations (up to 30 days)
  Thirty-day readmission and reoperations in relation to the index procedure
Functional outcomes-continence status | Post-operation 1/3/6/12 months
  Continence status after Foley catheter removed. Pad-free or one safe pad used are defined as continence intact. More than one pad used is defined as post-operative incontinence.
Functional outcomes-continence (pad amount) | Post-operation 1/3/6/12 months
  pads used per day (for patients with incontinence)
Functional outcomes-continence (leak amount in gram) | Post-operation 1/3/6/12 months
  24hr total weight of pads (for patients with incontinence)
Functional outcomes-sexual function change (IIEF-5) | Baseline, Post-operation 1/3/6/12 months
  sexual function at baseline and 1/3/6/12 months with International Index of Erectile Function (IIEF-5), 0-25, higher score indicates better sexual function.
Oncologic outcomes-margin status (positive or negative) | when the pathology report is available (up to day 10)
  surgical margin status
Oncologic outcomes-biochemical recurrence | Post-operation 1/3/6/12 months
  biochemical recurrence (PSA level ng/ml)

CONTACTS AND LOCATIONS:
Overall Officials: Chun-Te Wu, Professor, MD, PhD, Principal Investigator — Chang Gung Memorial Hospital at Keelung
Locations (1):
- Chang Gung Memorial Hospital, Taoyuan, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lin PH, Wang HJ, Kan HC, Pang ST, Yu KJ, Wu CT. Comparable oncological and functional outcomes of robot-assisted radical prostatectomy with conventional anterior approach and Hood technique using DAVINCI SP system. Sci Rep. 2025 Nov 28;15(1):45652. doi: 10.1038/s41598-025-30245-5. PMID 41315721